CLINICAL TRIAL: NCT07048782
Title: Development and Validation of a Risk Prediction Model for Postoperative Visceral Pain in Abdominal Surgery Patients
Status: Not yet recruiting | Type: Observational
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: vpclinicaltrial1
Record Dates: First submitted 2025-06-15; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Postoperative Visceral Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective Cohort: This cohort includes 1000 patients whose data were collected retrospectively from existing medical records. No additional follow-up is planned.
  Interventions: Other: Observational assessment of clinical outcomes
- Prospective Cohort: This cohort includes 135 patients enrolled prospectively and followed for 2 days to collect outcomes and relevant clinical data.
  Interventions: Other: Observational assessment of clinical outcomes

INTERVENTIONS:
Other: Observational assessment of clinical outcomes — This is a non-interventional observational study. No treatment or behavioral intervention is administered.

SUMMARY:
This study aims to investigate the factors influencing the risk of postoperative visceral pain in patients undergoing abdominal surgery. The goal is to develop and validate a predictive model for assessing the risk of postoperative visceral pain, in order to guide individualized preoperative interventions and pain management strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective abdominal surgery under general anesthesia (including gynecological procedures and general surgery such as gastrointestinal, hepatobiliary, etc.);
* Aged between 18 and 70 years;
* Classified as American Society of Anesthesiologists (ASA) physical status II-III;
* Expected surgery duration ≥ 2 hours.

Exclusion Criteria:

* History of previous abdominal surgery;
* Diagnosed with chronic pain;
* Long-term use of analgesics or other psychotropic medications;
* Preoperative emergency condition;
* Presence of severe comorbidities involving major organ systems;
* Failure to complete postoperative pain follow-up.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 to 70 years who are scheduled to undergo elective abdominal surgery under general anesthesia (including gynecological and general surgeries such as gastrointestinal and hepatobiliary procedures), with an ASA physical status of II to III, and an expected surgery duration of 2 hours or more.
Sampling Method: Non-Probability Sample
Enrollment: 1135 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity after surgery | From end of surgery to 48 hours postoperatively
  Pain intensity will be recorded at 6, 12, 24, and 48 hours after surgery. At each time point, the Numerical Rating Scale (NRS) pain score will be assessed both at rest and during coughing. Pain intensity was assessed using number rating scale (0-10, higher score represents worse pain intensity)

SECONDARY OUTCOMES:
Postoperative Length of Hospital Stay | From end of surgery to hospital discharge (up to 30 days)
  The total time from the end of surgery to hospital discharge will be recorded for each patient. The duration will be measured in days (d) and used to assess postoperative recovery.
Postoperative Analgesic Use | From end of surgery to hospital discharge (up to 30 days)
  Detailed records will be kept of the types of analgesics administered postoperatively, the total dosage of each drug, and the frequency of use per day. This measure will help assess pain management and medication requirements after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Guangyou Duan, PhD, Principal Investigator — The Second Affiliated Hospital, Chongqing Medical University
Locations (1):
- Department of Anesthesiology, The Second Affiliated Hospital, Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data for this study is available from the sponsor on reasonable request through email.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Five years after the study